CLINICAL TRIAL: NCT03977103
Title: Antileukemic Activity of Allogeneic Hematopoietic Stem Cell Transplantation With Fractionated Total Body Irradiation or Total Marrow and Lymph Node Irradiation Followed by Adoptive Immunotherapy With Regulatory and Conventional T Cells
Brief Title: Irradiation-based Myeloablative Conditioning Followed by Treg/Tcon Immunotherapy in HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Andrea Velardi, Full Professor, University Of Perugia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02/14
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Myeloproliferative Disorders; Lymphoma; Multiple Myeloma; Other Hematologic Malignant Neoplasms
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myeloproliferative Disorders; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High dose irradiation conditioning + Treg/Tcon (Experimental): High dose irradiation based conditioning regimens followed by infusion of donor regulatory and conventional T cells and purified CD34+ hematopoietic stem cell transplantation
  Interventions: Biological: High dose irradiation conditioning + Treg/Tcon

INTERVENTIONS:
Biological: High dose irradiation conditioning + Treg/Tcon — High dose irradiation based conditioning regimens followed by infusion of donor regulatory and conventional T cells and purified CD34+ hematopoietic stem cell transplantation

SUMMARY:
To evaluate if hyper-fractionated TBI or TMLI followed by Treg/Tcon adoptive immunotherapy improve cGvHD/disease free survival after allogeneic HSCT in patients affected by high-risk acute leukemias or other hematologic malignancy where HSCT is indicated.

DETAILED DESCRIPTION:
Improving cGvHD/disease free survival in patients with high-risk acute leukemias or other hematologic malignancy where HSCT is indicated with the use of a regulatory T cell based protocol. Hyper-fractionated Total Body Irradiation or Total Marrow and Lymphoid Irradiation based conditioning will be followed by the infusion of T regulatory and T conventional cell adoptive immunotherapy and a purified CD34+ hematopoietic stem cell graft. Incidence of Non Relapse Mortality, Relapse, acute Graft versus Host Disease, chronic Graft versus Host Disease, as well as probability of cGvHD/disease free survival will be assessed in patient subpopulations separated according to HLA-matching with the donor (HLA-matched HSCT and HLA-haploidentical HSCT) and type of disease (acute myeloid leukemia, acute lymphoid leukemia, lymphoma, multiple myeloma, myeloproliferative disease, and other).

ELIGIBILITY:
Inclusion Criteria:

* AML and ALL in complete remission and with high-risk of relapse
* AML and ALL primarily chemoresistant or relapsed;
* Chronic Myeloid Leukemia in accelerated or blastic phase;
* Patients affected by

  * Multiple myeloma,
  * Non Hodgkin lymphoma,
  * Hodgkin lymphoma,
  * Chronic myeloproliferative syndrome,
  * Chronic Lymphoid Leukemia,
  * Other Hematological malignancy at high-risk of relapse or detectable disease and where a HSCT is indicated.
* Age <75 years
* ECOG ≤ 2
* Acceptable lung, liver, kidney, and heart function and absence of relevant psichiatric diseases
* Signature of the informed consent

Exclusion Criteria:

* Age >75 years
* ECOG > 2
* Not acceptable lung, liver, kidney, and heart function and presence of relevant psichiatric diseases
* Pregnancy
* No signature of the informed consent

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-02; Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
chronic GvHD/relapse-free survival | 2 years
  To evaluate if irradiation based myeloablative conditioning followed by Treg/Tcon adoptive immunotherapy improve chronic GvHD/relapse-free survival (GRFS) after allogeneic HSCT in patients affected by acute leukemias or other hematologic malignancies where HSCT is indicated. GRFS will be assessed in subgroups of patients separated according to HLA-matching with the donor and type of disease (acute myeloid lekemia, acute lymphoid leukemia, other)

SECONDARY OUTCOMES:
full donor-type engraftment | 30 days
  neutrophil and platelet engraftment measured by neutrophil counts >500/mmc for 3 consecutive days and platelets count >20000/mmc with 7 consecutive without platelet transfusion

OTHER OUTCOMES:
cumulative incidence of grades ≥ 2 acute GvHD | 6 months
  cumulative incidence of grades ≥ 2 acute GvHD according to NIH consesus criteria
cumulative incidence of extensive chronic GvHD | 2 years
  cumulative incidence of extensive chronic GvHD according to revised NIH consesus criteria (Jagasia et al. BBMT 2015)
cumulative incidence of non-relapse mortality | 2 years
  cumulative incidence of non-relapse mortality, defined as death by any cause in the absence of relapse, as competitive risk versus relapse
cumulative incidence of relapse | 2 years
  cumulative incidence of relapse, defined as disease recurrence according to marrow morphology, flow cytometry, cytogenetics, fluorescence in situ hybridization and/or polymerase chain reaction, as competitive risk versus non-relapse mortality

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Velardi, MD, PhD, Principal Investigator — University Of Perugia
Locations (1):
- University of Perugia, Perugia, PG, Italy

REFERENCES:
- [Background] Di Ianni M, Falzetti F, Carotti A, Terenzi A, Castellino F, Bonifacio E, Del Papa B, Zei T, Ostini RI, Cecchini D, Aloisi T, Perruccio K, Ruggeri L, Balucani C, Pierini A, Sportoletti P, Aristei C, Falini B, Reisner Y, Velardi A, Aversa F, Martelli MF. Tregs prevent GVHD and promote immune reconstitution in HLA-haploidentical transplantation. Blood. 2011 Apr 7;117(14):3921-8. doi: 10.1182/blood-2010-10-311894. Epub 2011 Feb 3. PMID 21292771
- [Background] Martelli MF, Di Ianni M, Ruggeri L, Falzetti F, Carotti A, Terenzi A, Pierini A, Massei MS, Amico L, Urbani E, Del Papa B, Zei T, Iacucci Ostini R, Cecchini D, Tognellini R, Reisner Y, Aversa F, Falini B, Velardi A. HLA-haploidentical transplantation with regulatory and conventional T-cell adoptive immunotherapy prevents acute leukemia relapse. Blood. 2014 Jul 24;124(4):638-44. doi: 10.1182/blood-2014-03-564401. Epub 2014 Jun 12. PMID 24923299
- [Derived] Pierini A, Ruggeri L, Carotti A, Falzetti F, Saldi S, Terenzi A, Zucchetti C, Ingrosso G, Zei T, Iacucci Ostini R, Piccinelli S, Bonato S, Tricarico S, Mancusi A, Ciardelli S, Limongello R, Merluzzi M, Di Ianni M, Tognellini R, Minelli O, Mecucci C, Martelli MP, Falini B, Martelli MF, Aristei C, Velardi A. Haploidentical age-adapted myeloablative transplant and regulatory and effector T cells for acute myeloid leukemia. Blood Adv. 2021 Mar 9;5(5):1199-1208. doi: 10.1182/bloodadvances.2020003739. PMID 33646302